## Pain, Agitation and Delirium (PAD) Protocol in the Duke CICU

NCT02903407

**April 30, 2020** 

## **Statistical Analysis Plan**

Baseline patient characteristics, including age, sex, race, BMI and baseline ejection fraction for the participants will be described, both for the overall cohort and by randomization group.

The primary outcome measure – ICU length of stay – will be described for the overall population and by randomization group. Each of the secondary outcomes will also be described for the entire cohort and each group. Categorical variables will be presented using percentages and continuous variables using medians (25th and 75th percentiles). Given the small number of patients in the study, only descriptive results will be completed.